CLINICAL TRIAL: NCT02018614
Title: INTERNATIONAL VALIDATION STUDY OF THE ALGOPLUS SCALE IN FIVE LANGUAGES
Acronym: ALGOPLUS LE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr M Fisher Dr. Ulrike Bornschlegel (Unknown); Dr M Schuler (Unknown); Dr Pat Schofield (Unknown); Dr D Lussier (Unknown); Dr S Gibson (Unknown); Dr Joan ESPAULELLA PANICOT (Unknown); Dr Joan Manuel PEREZ CASTEJON (Unknown); Gambassi, Giovanni, M.D. (Individual); Dr Patrizio ODETTI (Unknown); Dr Fiametta MONACELLI (Unknown); University Hospital, Grenoble (Other); Dr Hirondina GUARDA, Dr Sónia SANTOS (Unknown); Dr Gisèle PICKERING (Unknown); Dr Valérie LEGOUT (Unknown); Dr Patrice Rat (Unknown); Dr Bernard WARY (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0172
Record Dates: First submitted 2013-12-06; First posted 2013-12-23 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pain; Elderly; Communication Disorders
Keywords: Pain; elderly; aged 65 or above 65; communication disorders; Algoplus® scale
MeSH Terms: conditions — Pain; Communication Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- testretest relaibility: Data from a sample of 50 patients will be used to explore the test-retest reliability of the scale administered by the same trained clinician, on two occasions four hours apart, without any treatment in between. The ALGOPLUS® scores obtained from the patients at a time t will be compared with their (t + 4 hours) scores to assess test-retest reliability
  Interventions: Other: algoplus
- statistical test: For a sample of at least 50 patients, two physicians trained for the use of ALGOPLUS, will assess pain independently. A statistical test will be used to compare the results for the inter-rater reliability
  Interventions: Other: algoplus

INTERVENTIONS:
Other: algoplus

SUMMARY:
Acute pain is responsible for unnecessary suffering. Among elderly patients, acute pain is frequent and underestimated, especially when these patients have cognitive disorders. The expression of pain is then modified and the conventional tools for evaluating pain cannot be used. Thus the existence of pain must be detected on the basis of a behavioural assessment.

It is nonetheless necessary to have the assistance of standardised and validated tools. In France, the Doloplus Group has proposed a scale called Doloplus, validated in January 1999, and is now proposing a new scale for acute pain, Algoplus that has been validated in French (4). Doloplus has been recently translated and validated in 5 languages and an identical methodology will be used in this protocol.

Internationally, although several teams are working on the development of scales that can be used for non-communicating elderly subjects, there is as yet no validated tool for acute pain assessment.

Considering 1- the lack of tools at an international level and 2- the frequent request from many practitioners worldwide, the Doloplus group has offered to validate the Algoplus® scale in 5 foreign languages, English, German, Spanish, Italian, Portuguese. A rigorous methodology with the help of a statistician will be used in this validation process.

DETAILED DESCRIPTION:
50 patients per language will be explored : t1 = time t Physician M Physician N t2 = time t+4 hours Physician M

The methodology of the validation of our translation procedure consists of studying the reliability of the scale in two major steps:

* Data from a sample of 50 patients will be used to explore the test-retest reliability of the scale administered by the same trained clinician, on two occasions four hours apart, without any treatment in between. The ALGOPLUS® scores obtained from the patients at a time t will be compared with their (t + 4 hours) scores to assess test-retest reliability.
* For a sample of at least 50 patients, two physicians trained for the use of ALGOPLUS, will assess pain independently. A statistical test will be used to compare the results for the inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

* - males or females aged 65 or above 65, with communication disorders
* with or without suspected acute pain

Exclusion Criteria:

* - are too agitated,
* have acute pain needing immediate pain management,
* change of treatment between the two evaluations ( t and t+4 hours ),
* refuse to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Inter-rater scale and intra-rater comparisons of the filled Algoplus® scale. | at time 1 (Physician N and M), at time 2 (t+4 hours) by physician M.
  The scale includes five items (facial expression, sight expression, complaints, bodily attitudes and finally the general behaviour).. The presence of one behaviour in each of the items is sufficient to score "yes" for the item under consideration.
  Each item marked "yes" is scored one point and the sum of the items provides a total score out of five

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France